CLINICAL TRIAL: NCT06674733
Title: Evaluation of the Efficacy of Botulinum Toxin and Marjoram Oil Applications in Sleep Bruxism
Brief Title: Efficacy of Botulinum Toxin and Marjoram Oil Applications in Bruxism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13.02.2024-E.140948
Record Dates: First submitted 2024-10-30; First posted 2024-11-05 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Bruxism, Sleep
Keywords: Bruxism; Botox; Origanum Majorana; Ultrasonography
MeSH Terms: conditions — Sleep Bruxism; Bruxism | interventions — Aromatherapy; Time-Lapse Imaging

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botox group (Active Comparator): Group 1 will consist of patients with bruxism complaints who are indicated for botox treatment and will receive BTX-A.
  Interventions: Procedure: Botox administration; Procedure: Clinical evaluation; Procedure: Imaging Time
- aromatherapy group (Active Comparator): Group 2 will consist of patients with bruxism complaints and will receive Origanum Majorana (marjoram oil)
  Interventions: Procedure: Aromatherapy; Procedure: Clinical evaluation; Procedure: Imaging Time

INTERVENTIONS:
Procedure: Botox administration — Treatment for bruxism
  Arms: Botox group
Procedure: Aromatherapy — treatment for stress-bruxism
  Arms: aromatherapy group
Procedure: Clinical evaluation — Before the procedure, and at 1 month and 3 months after the procedure, the Fonseca questionnaire, symptom assessment questionnaire, and Basic Scale on Insomnia Complaint and Quality of Sleep (BaSIQS) will be administered. At the 1st month and 3rd month, Subject Global Aesthetic Improvement Scale (GAIS), and satisfaction questionnaire will be administered
Procedure: Imaging Time — Ultrasonography and shear wave elastography examination will be performed before the procedure, one month after, and three months after the procedure.

SUMMARY:
Objective: Bruxism is defined as clenching or grinding teeth unconsciously. It can be categorized under two subheadings: sleep and awake bruxism. This study aims to investigate the effectiveness of botox applications, a current approach in the treatment of sleep bruxism, and to evaluate the effectiveness of alternative therapies like aromatherapeutic oils. The study will compare and assess the efficacy of these methods.

Materials and Methods: This prospective study will be conducted between March 2024 and January 2025 at Bezmialem Vakıf University, Faculty of Dentistry, Department of Oral and Maxillofacial Radiology, with patients aged between 18 and 60 who have presented complaints of clenching/grinding teeth, sleep bruxism, jaw, neck, or face pain, and insomnia. The patients diagnosed with sleep bruxism will be divided into two groups, each consisting of 15 patients. The first group will include 15 patients with sleep bruxism who will receive botulinum toxin-A (BTX-A) injections, and the second group will consist of 15 patients who will use marjoram oil as an alternative treatment. Ultrasound imaging will assess the thickness and stiffness of the masseter muscle before treatment, and at 1 and 3 months post-treatment. Clinical evaluations will also be performed before treatment, and at 1 and 3 months post-treatment using scoring systems.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported teeth clenching or grinding
2. Tenderness or fatigue in the masticatory muscles upon palpation
3. Increased morning muscle pain
4. Localized myofascial pain in the jaw, face, or neck region
5. Irregular or excessive enamel wear consistent with bruxism
6. Grinding sounds during sleep confirmed by a partner
7. Morning jaw muscle stiffness and spasms causing sleep disturbances
8. Individuals older than 18 years,
9. Individuals younger than 60 years,
10. Provided informed voluntary consent

Exclusion Criteria:

1. Botulinum toxin injection into the masseter muscle within the last 6 months
2. Use of night guards
3. Pathology or history of surgery involving the masseter muscle or parotid gland
4. Benign or malignant tumors in the mandibular region
5. History of alcohol or substance abuse
6. Age below 18 or above 60
7. Pregnancy, postpartum period, or breastfeeding
8. Infection or dermatological lesions at the injection site
9. Diagnosis of chronic obstructive pulmonary disease (COPD) or asthma
10. Known allergy or skin reaction to botulinum toxin A or essential oils used in aromatherapy
11. Use of muscle relaxants or other medications that may affect muscle function

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-10-11 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Evaluation of Changes in Bruxism Symptoms with scales (The Fonseca Anamnestic Index) | From enrollment to the 3-month follow-up after the procedure.
  It is an index ranging from 0 to 100 for classifying the severity of TMD. A score of 0-15 indicates no TMD, 20-40 indicates mild TMD, 25-65 indicates moderate TMD, and 70-100 indicates severe TMD.
USG examination | From enrollment to the 3-month follow-up after the procedure.
Evaluation of Changes in Bruxism Symptoms with scales (Subject Global Aesthetic Improvement Scale) | From enrollment to the 3-month follow-up after the procedure.
  It is a scoring system between 0 and 4. A score of 0 indicates that the condition is worse than before the procedure, while a score of 4 indicates an ideal outcome.
Evaluation of Changes in Bruxism Symptoms with scales (Basic Scale on Insomnia Complaint and Quality of Sleep) | From enrollment to the 3-month follow-up after the procedure.
  It is a scoring system between 0 and 28. A score of 0 indicates no problems related to sleep, while a score of 28 represents severe insomnia complaints and poor sleep quality.
Satisfaction Survey | From enrollment to the 3-month follow-up after the procedure.
  It is a scoring system between 1 and 5. A score of 1 indicates complete dissatisfaction, while a score of 5 indicates a high level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Elifhan Alagoz, Asst. Prof., Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The purpose of this study was to evaluate the efficacy and safety of onabotulinumtoxin A and Chinese botulinum toxin type A (CBA) for masseter reduction using elastography and electromyographic measurement. — https://pubmed.ncbi.nlm.nih.gov/35758504/
- See also: This study aimed to evaluate the correlation between the changes in masseter muscle thickness and clenching habits in bruxism patients treated with BT-A. — https://pubmed.ncbi.nlm.nih.gov/37180633/
- See also: This study aimed to investigate the effect of inhalation of marjoram essential oil at work on the stress and anxiety levels of nurses in a COVID-19 ICU. — https://pubmed.ncbi.nlm.nih.gov/38045619/